CLINICAL TRIAL: NCT03040297
Title: Effect of Parallel Oxygen Delivery Through a Tracheal Gas Insufflation (TGI) and a T-piece on Blood Gases and Respiratory Rate in ICU Tracheostomized Patients as an Extra Supporting Method During Weaning From Mechanical Ventilation.
Brief Title: Effect of Parallel Oxygen Delivery Through a Tracheal Gas Insufflation (TGI) and a T-piece, on Blood Gases and Respiratory Rate, in ICU Tracheostomized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Konstantinos Grigoriadis, Physical Therapist, Attikon Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 13.4.4.25/05/16
Record Dates: First submitted 2017-01-27; First posted 2017-02-02 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Resp Gas Exchange Disorder Nos
Keywords: Weaning from mechanical ventilation; tracheostomized patients; Tracheal gas insufflation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TGI 6 L/min (Active Comparator): Tracheal gas insufflation 6 L/min
  Interventions: Device: Tracheal gas insufflation 6 L/min
- TGI 11 L/min (Active Comparator): Tracheal gas insufflation 11 L/min
  Interventions: Device: Tracheal gas insufflation 11 L/min
- TGI 0 L/min (Active Comparator): Tracheal gas insufflation catheter, without gas flow
  Interventions: Device: Tracheal gas insufflation catheter, without gas flow

INTERVENTIONS:
Device: Tracheal gas insufflation 6 L/min — Endotracheal flow (6 L/min) of respiratory gases with standard FiO2
  Arms: TGI 6 L/min
Device: Tracheal gas insufflation 11 L/min — Endotracheal flow (11 L/min) of respiratory gases with standard FiO2
  Arms: TGI 11 L/min
Device: Tracheal gas insufflation catheter, without gas flow — Tracheal gas insufflation catheter, without gas flow
  Arms: TGI 0 L/min

SUMMARY:
The study investigates if there are benefits (better oxygenation, minimized work of breath) from the parallel oxygenation with Tracheal Gas Insufflation and T-piece, in order to provide respiratory support in tracheostomized patients and avoid mechanical ventilation.

DETAILED DESCRIPTION:
The tracheal insufflation (TGI) of respiratory gasses near to carina is a technique who designed for the removement of exhaled carbon dioxide from the dead space of the lung. In order to investigate the utility of this technique on weaning of mechanical ventilation 11 tracheostomized patients on T-piece were recruited, with stable blood gasses more than 24 hours.

A TGI catheter enters the trachea through a new opened hole on the top of T-piece and then passes through the tracheostomy tube to inside of the trachea and then stops one centimeter before the carina. Patients received two parallel administered respiratory gases with the same fraction of inspired oxygen (FiO2), through a T-piece and an endotracheal catheter, with flows 6 Liters Per Minute (L/min) and 11 L/min, while continuously monitored by impedance tomography device (ΕΙΤ). ΕΙΤ is a noninvasive imaging technique for monitoring in real time the lung volumes and the regional lung ventilation without ionizing radiation.

The basic hypothesis of the study is if there are benefits (better oxygenation, minimized work of breath) from the parallel oxygenation with Tracheal Gas Insufflation and T-piece, in order to provide respiratory support in tracheostomized patients and avoid mechanical ventilation.

The randomization of the study was achieved using sealed envelopes method and associated with the flow to be first (6L/min or 11L/min) via Tracheal Gas Insufflation Catheter (6 envelopes with the inscription 6 L/min on the inner side and 6 envelopes with the inscription 6 L/min on the inner side 11 L/min)

Τhe investigators tested the differences on partial pressure of oxygen (PaO2), respiratory rate and end expiratory impedance:

1. Before gasses supply via TGI
2. During 6L/min
3. During 11L/min
4. And finally with no gasses supply via TGI

Additionally the following were monitored:

* Heart rate
* Systolic and diastolic blood pressure
* Oxygen saturation as disturbing factors and,
* potential of hydrogen (pH)
* PaCO2
* hydrogen carbonate (-HCO3) for the monitoring of the acid-base balance of the patient during procedure.

ELIGIBILITY:
Inclusion Criteria:

* Tracheostomized haemodynamically stable patients, without the need of vasopressors or inotrope medications, without symptoms of pulmonary edema, or interstitial lung diseases.

Stable blood gasses (no bigger changes than 15-20% in Oxygen and Carbon dioxide during last 24 hours)

Exclusion Criteria:

* Peripheral body temperature < 38 C, White blood cells (WBCs) < 15 x 109/L
* Respiratory rate >35
* Paradoxical breathing
* Abdominal muscle recruitment
* Dyspnoea, SaO2 < 94, without evidence of angina, cyanosis or arrhythmia.
* Chest circumferences no bigger than 110 cm (for the larger belt of impedance tomograph)

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-11; Primary Completion 2017-01 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Respiratory Rate | 60 minutes
  Respiratory cycles per minute at flows: 0, 6, 11, 0 L/min
partial pressure of oxygen (PaO2) | 60 minutes
  Arterial blood oxygen tension at flows: 0, 6, 11,0 L/min
End respiratory lung impedance differences | 60 minutes
  End respiratory lung impedance differences at flows: 0, 6, 11, 0 L/min

SECONDARY OUTCOMES:
Heart Rate | 60 minutes
  Heart beats per minute at flows: 0, 6, 11, 0 L/min
Systolic blood pressure | 60 minutes
  Systolic blood pressure (mmHg) at flows: 0, 6, 11, 0 L/min
Diastolic blood pressure | 60 minutes
  Diastolic blood pressure (mmHg) at flows: 0, 6, 11, 0 L/min
Oxygen saturation (SaO2) | 60 minutes
  Oxygen saturation (%) at flows: 0, 6, 11, 0 L/min

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos E Grigoriadis, Pt, MSc, Principal Investigator — National and Kapodistrian University of Athens; Iraklis Tsagaris, MD. PhD, Study Chair — National and Kapodistrian University of Athens; Antonia D Koutsoukou, MD, PhD, Study Chair — National and Kapodistrian University of Athens; Eirini P Grammatopoulou, PT, PhD, Study Chair — Technological Educational Institution of Athens; Anna K Grigoriadou, PT, Study Chair — Lamia University of Applied Sciences; Apostolos E Armaganidis, Study Director — National and Kapodistrian University of Athens
Locations (1):
- Attikon University Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knebel AR. When weaning from mechanical ventilation fails. Am J Crit Care. 1992 Nov;1(3):19-29; quiz 30-1. PMID 1307903
- [Background] Durbin CG Jr. Tracheostomy: why, when, and how? Respir Care. 2010 Aug;55(8):1056-68. PMID 20667153
- [Background] Blanch LL. Clinical studies of tracheal gas insufflation. Respir Care. 2001 Feb;46(2):158-66. PMID 11175244
- [Background] Hoffman LA, Tasota FJ, Delgado E, Zullo TG, Pinsky MR. Effect of tracheal gas insufflation during weaning from prolonged mechanical ventilation: a preliminary study. Am J Crit Care. 2003 Jan;12(1):31-9. PMID 12526235
- [Background] Hess DR, Gillette MA. Tracheal gas insufflation and related techniques to introduce gas flow into the trachea. Respir Care. 2001 Feb;46(2):119-29. PMID 11175241
- [Background] Nahum A. Animal and lung model studies of tracheal gas insufflation. Respir Care. 2001 Feb;46(2):149-57. PMID 11175243
- [Background] Kacmarek RM. Complications of tracheal gas insufflation. Respir Care. 2001 Feb;46(2):167-76. PMID 11175245